CLINICAL TRIAL: NCT02986347
Title: Surgical Treatment of Carpal Tunnel Syndrome: Local Anesthesia With Epinephrine x Intravenous Regional Anesthesia. Randomized Clinical Trial.
Brief Title: Surgical Treatment of Carpal Tunnel Syndrome: Local Anesthesia With Epinephrine x Intravenous Regional Anesthesia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Alvorada (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, João Carlos Belloti, PhD, Hospital Alvorada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HAMAO01
Record Dates: First submitted 2016-11-11; First posted 2016-12-08 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Carpal Tunnel Syndrome; Anesthesia
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Anesthesia, Local; Epinephrine

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous regional anesthesia (Bier) (Active Comparator): The anesthetic technique described by Bier will be done by the anesthesiologist. The following steps were followed: 1)Placement double tourniquet on the proximal portion of the arm 2)Asepsis and antisepsis of the operative limb 3)Puncture and venous catheterization most distal in the limb 4)Elevation of limb for 1 to 2 minutes, next the limb will be spirally wrapped with Esmarch from the distal to proximal 5)The proximal cuff will be inflated 6)Withdrawal of Esmarch and injection of 40ml of lidocaine without epinephrine at 0.5% 7)Removal the canula until the distal cuff is inflated and the proximal cuff is emptied 8)Removal of the club must be done after the surgery, at least 40 minutes after the injection of the anesthetic.
  Interventions: Procedure: Intravenous regional anesthesia (Bier)
- Local anesthesia with adrenaline (Active Comparator): Patients will be anesthetized by surgeons, who are familiar with the technique described by Lalonde. Around thirty minutes before surgery, will be infused with 20 ml of an anesthetic solution. The infiltrated solution is composed of 1% lidocaine with epinephrine in 1: 100,000. Initially 10 mL of the solution will be applied slowly in the flexion fold region of the wrist just below the skin and subfascial plane. The needle is moved slowly. The needle is then redirected to the radial side of the proximal palmar region for infiltration of another 2-3 mL of the subcutaneous solution. The remaining 7-8mL in the subdermal plane and anterior to the transverse carpal ligament.
  Interventions: Procedure: Local anesthesia with adrenaline

INTERVENTIONS:
Procedure: Intravenous regional anesthesia (Bier) — Intravenous regional anesthesia (Bier Technique)
  Arms: Intravenous regional anesthesia (Bier)
Procedure: Local anesthesia with adrenaline — local anesthesia with adrenaline without limber garroting (Lalonde Technique)
  Arms: Local anesthesia with adrenaline

SUMMARY:
The anesthetic technique of choice for surgical treatment of CTS varies among surgeons. In the last decade some studies have described the performance of this surgery using local anesthesia with adrenaline without the necessity of sedation or the use of pneumatic garrote, having good effectiveness and substantial reduction of costs. However there is need for studies with an appropriate design and methodology to evaluate the actual effectiveness of this kind of anesthesia for the surgical treatment of CTS.

Objective: To evaluate the effectiveness and cost of open surgery for CTS in a randomized trial comparing two anesthesia methods: intravenous regional anesthesia (Bier) and local anesthesia with adrenaline without limb garroting (Lalondi).

Methods: This study was developed in the Group of Hand Surgery and Upper Limb; Department of Orthopedics and Traumatology, Federal University of São Paulo, UNIFESP / EPM with co-participation of the Hand Surgery and Microsurgery Department of Hospital Alvorada. This study will be a Randomized Clinical Trial. The previous calculation of the sample resulted in 78 patients. The following primary outcomes will be assessed: Pain through visual analogue scale (VAS). Costs: Costs related to anesthetic and surgical procedures will be recorded. The secondary outcomes will be: Use of Analgesics, Anxiety and Depression through the HADS (Hospital Anxiety and Depression Scale) scale. Quality of life through the Boston Carpal Tunnel Syndrome Questionnaire (BCTQ). Remission of paresthesia after surgical intervention, complications and failures.

DETAILED DESCRIPTION:
Surgical treatment of CTS is most often performed under hospital conditions, with the use of anesthesia. The anesthetic technique of choice varies among surgeons. In the last decade some studies have described the performance of this surgery using local anesthesia with adrenaline without the necessity of sedation or the use of pneumatic garrote, having good effectiveness and substantial reduction of costs for the procedure with this anesthetic method. However, when we evaluated the level and strength of the evidence from these studies, we notice that there is a need for studies with an appropriate design and methodology to evaluate the actual effectiveness of this kind of anesthesia for the surgical treatment of CTS.

Objective: To evaluate the effectiveness of open surgery for CTS in a randomized trial comparing two anesthesia methods: intravenous regional anesthesia (Bier) and local anesthesia with adrenaline without limb garroting (Lalondi).

Methods: This study was developed in the Group of Hand Surgery and Upper Limb; Department of Orthopedics and Traumatology, Federal University of São Paulo, UNIFESP / EPM with co-participation of the Hand Surgery and Microsurgery Department of the Medical Residency Service in Hand Surgery of Hospital Alvorada. This study will be a Randomized Clinical Trial. The previous calculation of the sample resulted in the need for total inclusion of 35 patients in each group, total of 70 patients, considering a loss of 10% during follow-up we will include 78 patients. The following primary outcomes will be assessed: Pain through visual analogue scale (VAS), that, will be measured in the pre-operative, transoperatory, immediate postoperative, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours after surgery. Costs: Costs related to anesthetic and surgical procedures will be recorded. The secondary outcomes will be: Use of Analgesics, Anxiety and Depression through the HADS (Hospital Anxiety and Depression Scale) scale. Quality of life through the Boston Carpal Tunnel Syndrome Questionnaire (BCTQ). Remission of paresthesia after surgical intervention, complications and failures.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age, with idiopathic Carpal Tunnel Syndrome with indication for surgery due to failure of conservative treatment for at least three months or that presented at the initial diagnosis with motor impairment detected by clinical examination (hypotrophy) and/or by electromyography (ENMG) examination.
* The diagnosis of CTS will be made through the clinical evaluation in which CTS patients will be considered, those who present at least four of the clinical criteria proposed and proven by the electromyography examination.

Clinical Criteria for CTS - (At least 4 criteria will be required for clinical confirmation of the diagnosis)

1. Paresthesia in the territory of the median nerve
2. Night paresthesia of the hand
3. Decreased strength with hypotrophy of the musculature tenar
4. Positive tinnitus sign on the wrist
5. Positive Phalen test
6. Loss of 2-point discrimination in the region innervated by the median nerve

   * Patients who agree to participate, after having been adequately informed about the nature of the study, and have reading and signed the informed consent form.

Exclusion Criteria:

* Patients with prior history of cervical spine diseases (radiculopathies, arthrosis),
* Pregnant women and puerperal women,
* Patients with sequelae of previous wrist and hand surgeries,
* Other upper limb compressive syndromes and scapular girdles will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-05-27 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change in pain through Pain visual analogue scale | Before the treatment and after the treatment (intraoperative and after the treatment:immediate postoperative, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours after the end of surgery.
  Pain measurement through visual analog scale

SECONDARY OUTCOMES:
The total costs of carpal tunnel syndrome surgical treatment will be tracked over the duration of the study to determine the cost-effectiveness of providing a Local Anesthesia With Epinephrine versus a Intravenous Regional Anesthesia. | 3 months
  The following costs related to anesthetic and surgical procedures will be computed:
  * consumer material used in the anesthetic and surgical procedure
  * medical and paramedical staff
  * time of use of the surgical rooms for postoperative recovery
  * length of hospital stay
  * medicines used up to one postoperative week
  * necessary costs for the treatment of possible complications
Change of the Boston Carpal Tunnel Questionnaire (BCTQ) | preoperatively and 12 weeks post-operation
  Patients in the study group will respond to Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) translated and validated for Portuguese preoperative (after initial clinical evaluation) and postoperative (3th month PO). It is a disease specific questionnaire, self-administered, and evaluates the severity of the symptoms and functional status of patients with CTS. The BCTQ assesses the symptoms and the severity, frequency, time and type. The functional degree of scale evaluates how the syndrome affects daily life. Issues relating to the severity scale are composed of 11 questions. Each question has five answers, placed in order of increasing severity of symptoms. The issues relating to the functional status are composed of 8 questions, each of which corresponds to a functional activity. Each activity has a 5-degree-answer of difficulty progressively worsening.
Hospital Anxiety and Depression Scale (HADS) | preoperatively and 12 weeks post-operation
  Hospital Anxiety and Depression Scale (HADS) questionnaire. The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression complains. Patients were defined as having anxiety or depression or both if the score was 8 or more in the corresponding subscale.
Remission or not of paresthesia until the third month | preoperatively and 12 weeks post-operation
  The absence of paresthesia reported by the patient after surgery will be considered as "cure". The not regression paresthesia referred by patients in this period will be considered as non-healing.
Record and evaluate all complications associated with the surgical procedure | 12 weeks post-operation
  Complications rate of surgical and anesthesic procedures in patients with CTS

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Okamura, MD, Principal Investigator — Hospital Alvorada de Moema
Locations (1):
- Aldo Okamura, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mckee DE, Lalonde DH, Thoma A, Dickson L. Achieving the optimal epinephrine effect in wide awake hand surgery using local anesthesia without a tourniquet. Hand (N Y). 2015 Dec;10(4):613-5. doi: 10.1007/s11552-015-9759-6. Epub 2015 Apr 14. PMID 26568713
- [Background] Davison PG, Cobb T, Lalonde DH. The patient's perspective on carpal tunnel surgery related to the type of anesthesia: a prospective cohort study. Hand (N Y). 2013 Mar;8(1):47-53. doi: 10.1007/s11552-012-9474-5. PMID 24426892
- [Background] Lalonde D, Bell M, Benoit P, Sparkes G, Denkler K, Chang P. A multicenter prospective study of 3,110 consecutive cases of elective epinephrine use in the fingers and hand: the Dalhousie Project clinical phase. J Hand Surg Am. 2005 Sep;30(5):1061-7. doi: 10.1016/j.jhsa.2005.05.006. PMID 16182068
- [Background] Levine DW, Simmons BP, Koris MJ, Daltroy LH, Hohl GG, Fossel AH, Katz JN. A self-administered questionnaire for the assessment of severity of symptoms and functional status in carpal tunnel syndrome. J Bone Joint Surg Am. 1993 Nov;75(11):1585-92. doi: 10.2106/00004623-199311000-00002. PMID 8245050
- [Background] Leblanc MR, Lalonde J, Lalonde DH. A detailed cost and efficiency analysis of performing carpal tunnel surgery in the main operating room versus the ambulatory setting in Canada. Hand (N Y). 2007 Dec;2(4):173-8. doi: 10.1007/s11552-007-9043-5. Epub 2007 May 30. PMID 18780048
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Robles DS, Esteves S, Liça M, Lopes D, Lima S, Sousa C. Tratamento da síndrome do túnel cárpico:anestesia geral versus local?. Rev Port Ortop e Traum 23(3):217-224, 2015.
- [Derived] Okamura A, Moraes VY, Fernandes M, Raduan-Neto J, Belloti JC. WALANT versus intravenous regional anesthesia for carpal tunnel syndrome: a randomized clinical trial. Sao Paulo Med J. 2021 Oct 11;139(6):576-578. doi: 10.1590/1516-3180.2020.0583.R2.0904221. eCollection 2021. PMID 34644765